CLINICAL TRIAL: NCT04560283
Title: Randomized Clinical Trial to Assess the Efficacy and Safety of HYDEAL-D® Application in Promoting the Restoration of Sexual Function in the Postpartum Period
Brief Title: HYDEAL-D® Application for Promoting the Restoration of Sexual Function in the Postpartum Period
Acronym: HYDEAL-D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ospedale Policlinico San Martino (Other)
Responsible Party: Principal Investigator, Fabio Barra, Principal Investigator, Ospedale Policlinico San Martino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYDEAL-D-1-2016
Record Dates: First submitted 2020-09-12; First posted 2020-09-23 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Vagina; Anomaly; Puerperium; Disease; Sexual Dysfunction
Keywords: Puerperium
MeSH Terms: conditions — Congenital Abnormalities; Puerperal Disorders; Sexual Dysfunction, Physiological | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group receiving HYALOGYN® (Experimental)
  Interventions: Drug: Vaginal gel HYALOGYN®
- Control group undergoing expectant management (Placebo Comparator)
  Interventions: Behavioral: Expectant management

INTERVENTIONS:
Drug: Vaginal gel HYALOGYN® — Vaginal gel HYALOGYN® (HYDEAL-D® 2%; Fidia Farmaceutici, Abano Terme, Italy) every 3 days up for 12 consecutive weeks
  Arms: Experimental group receiving HYALOGYN®
Behavioral: Expectant management — Expectant management for 12 consecutive weeks
  Arms: Control group undergoing expectant management

SUMMARY:
During postpartum and lactation, vaginal epithelium tends to have an impaired degree of hydration and lubrication. This may lead to vaginal dryness, burning sensation dyspareunia or itching, which negatively affect the sexual function of puerperal women.

This study aimed to evaluate the efficacy of HYDEAL-D® vaginal gel (HYALOGYN®, Fidia Farmaceutici, Abano Terme, Italy) application on promoting the restoration of sexual function in the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* Women from 18 to 40 years old;
* Women in the puerperium period (after vaginal delivery or cesarean section);
* Women that are breast-feeding, that are not breast-feeding or that are breast-feeding partially;

Exclusion Criteria:

* Allergy to hyaluronic acid gel;
* Women non-Italian speaking;
* Women with signs of vaginal infection;
* Women with a history of cancer of any site with recent genital bleeding of unknown origin; and patients with acute hepatopathy, embolic disorders, severe primary disease of kidney;
* Women who are attending or have attended other clinical trials within previous two weeks;
* Women with mental disorder and no insight

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 25 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of sexual function by FSFI | At baseline; 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Barra, MD, Principal Investigator — Ospedale San Martino
Locations (1):
- Ospedale Policlinico San Martino, Genova, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gustavino C, Sala P, Cusini N, Gravina B, Ronzini C, Marcolin D, Vellone VG, Paudice M, Nappi R, Costantini S, Ferrero S, Barra F. Efficacy and safety of prolonged-release hyaluronic acid derivative vaginal application in the postpartum period: a prospective randomised clinical trial. Ann Med. 2021 Dec;53(1):1589-1597. doi: 10.1080/07853890.2021.1974083. PMID 34477473